CLINICAL TRIAL: NCT02627989
Title: An Observational Study Investigating the Treatment Satisfaction of Atopic Dermatitis Patients Who Have Switched to Ointment (W/O Emulsion) Formulation of Very Strong Class Topical Corticosteroids
Acronym: Ointment TS-AD
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18690
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2018-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — diflucortolone valerate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diflucortolone valerate (Nerisona/Texmeten): Adult patients with atopic dermatitis switching from diflucortolone-valerate fatty ointment to ointment (water/oil emulsion) during autumn/ winter (Nov to Feb) or spring/ summer (May to Aug)
  Interventions: Drug: Diflucortolone valerate (Nerisona); Drug: Diflucortolone valerate (Texmeten)

INTERVENTIONS:
Drug: Diflucortolone valerate (Nerisona) — Potency Class II (classified as Very Strong class in Japan) topical corticosteroids
Drug: Diflucortolone valerate (Texmeten) — Potency Class II (classified as Very Strong class in Japan) topical corticosteroids

SUMMARY:
This study intends to investigate patient satisfaction of treatment with Ointment (W/O emulsion) formulations of Potency Class II topical corticosteroids (TCs) for atopic dermatitis (AD) patients in Japan. Objectives include measuring patient satisfaction, treatment adherence, itchiness, and AD severity scores.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with a diagnosis of atopic dermatitis who are treated with Fatty Ointment Potency Class II (Very strong class) TCs
* Patients who are scheduled to change the formulation of the Potency Class II TC from Fatty Ointment to Ointment (Water in Oil; Water per Oil emulsion) as per investigator's routine treatment practice
* Patients who are aged over 20
* Patients who are able to understand and sign a written informed consent

Exclusion Criteria:

-Patients participating in an investigational program with interventions outside of routine clinical practice

* Patients with any contraindication to TCs
* Patients who are regarded as ineligible by the investigator
* Patients who are pregnant or breastfeeding
* For Period 2 (Spring-Summer), patients enrolled in the Period 1

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by the investigator who will also be the treating physician. As an observational study, only patients who the investigator plans on switching to the ointment (W/O emulsion) from fatty ointment formulation will be eligible to participate. Patients will be recruited for each seasonal phase and same patients may not necessarily be observed between the two seasonal phases.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction measured by Treatment Satisfaction Questionnaire for Medication (TSQM-9) | 10 months
  A Patient Reported Outcome questionnaire assessing treatment satisfaction by recalling the last 2-3 weeks of treatment

SECONDARY OUTCOMES:
Treatment adherence measured by Morisky Medication Adherence Scale (MMAS-8-Item) | 10 months
Itchiness according to Visual Analogue Scale (VAS) | 10 months
Severity Scoring of Atopic Dermatitis (SCORAD) | 10 months
Eczema Area and Severity Index (EASI) | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Tsu, Mie-ken, Japan